CLINICAL TRIAL: NCT03121053
Title: Preventing Contrast Induced Nephropathy After Transcatheter Aortic Valve Replacement
Acronym: PANTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Jan van der Heyden, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PANTER_V1.1
Record Dates: First submitted 2017-04-06; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Aortic Valve Disease; Chronic Kidney Disease; Contrast Induced Nephropathy; Acute Kidney Injury
Keywords: transcatheter aortic valve implantation; transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Disease; Renal Insufficiency, Chronic; Acute Kidney Injury | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium bicarbonate (Active Comparator): 250ml 1.4% sodium bicarbonate 1 h before TAVR
  Interventions: Drug: sodium bicarbonate
- hypotone saline (Active Comparator): 0.65% sodiumchloride 1 ml/kg/h for 12 h before and 12 h after TAVR
  Interventions: Drug: hypotone saline

INTERVENTIONS:
Drug: sodium bicarbonate
  Arms: sodium bicarbonate
Drug: hypotone saline
  Arms: hypotone saline

SUMMARY:
Chronic kidney disease (CKD) and (subsequent) acute kidney injury are frequent in patients undergoing transcatheter aortic valve implantation (TAVI). Moreover, these patients are easily hypervolemic and susceptible for cardiac decompensation. Prevention of contrast induced nephropathy (CIN) has not yet been studied in these patients, and evidence on different strategies is urgently needed. The objective of this study is to evaluate the efficacy of 250ml 1.4% sodium bicarbonate versus hypotone saline (0.65% sodiumchloride) hydration prior to TAVI in patients with CKD to prevent CIN.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent.
2. Patient is undergoing TAVI.
3. Patient has an estimated GFR <60ml/min/1.73m2.

Exclusion Criteria:

1. Patient has end-stage kidney disease requiring dialysis.
2. Emergent TAVI (planned before next working day).
3. Recent exposure to radiographic contrast agents (within 2 days prior to the TAVI).
4. Allergy to contrast agent.
5. Planned administration of dopamine, mannitol, fenoldopam or N-acetylcysteine during the intended time of the study.
6. Need for continuous hydration therapy (e.g. sepsis).
7. Multiple myeloma.
8. Contra-indication to sodium bicarbonate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Contrast induced nephropathy | Day 3
  CIN is defined as an increase in Scr >0.5 mg/dL or 25% within 72 hours
Acute heart failure due to volume expansion | Day 3

SECONDARY OUTCOMES:
Composite of CIN or acute heart failure | Day 3
Maximal relative change in serum creatinine | Day 3
Acute kidney injury | Day 3
  According to AKIN classification
Need for dialysis | Day 30
Need for blood transfusions | Day 3 and Day 30
Number of blood transfusions | Day 3 and Day 30
Length of hospital stay | Day 30
Recovery of renal function in CIN patients | Day 30
  Recovery defined as an increase in serum creatinine <25% or <44 μmol/L (0.5 mg/dL) measured at 1 month post-TAVI compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius hospital, Nieuwegein, Utrecht, Netherlands